CLINICAL TRIAL: NCT04479553
Title: Post-marketing Safety Surveillance of Qizhi Tongluo Capsules:a Registry Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhong Wang (Other)
Collaborators: Shanxi Zhendong Pharmacy Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: QZTL-V1.0
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Safety Surveillance; Adverse Drug Events; Adverse Drug Reactions; Severe Adverse Events; Severe Adverse Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — 1. The blood routine, urine routine, and stool routine before and after medication need to be obtained in the patients with adverse events
  2. The level of the liver functional indicators (including ALT,AST,ALP,TBIL,DBIL) the renal functional indicators (including BUN,SCr,UA) and the immune indicators (including IgA，IgE,the counts of T lymphocyte and B lymphocyte,CD3，CD4，CD8，CD20,serum histamine concentration,C3,C4) should be obtained in patients with serious adverse events and suspicious unexpected serious adverse reactions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qizhi Tongluo Capsules: Qizhi Tongluo Capsules will be given to the patients, and the investigators will record all the information including ADR, application of Qizhi Tongluo Capsules and the combined medications, etc.
  Interventions: Drug: Qizhi Tongluo Capsules

INTERVENTIONS:
Drug: Qizhi Tongluo Capsules — Qizhi Tongluo Capsule, a Chinese patent medicine composed of 26 Chinese herbs, has been approved by China Food and Drug Administration for treating recovery period of ischemic stroke (drug approval numbers: B20171001).

SUMMARY:
This registry aims to monitor the safety of Qizhi Tongluo Capsules and to identify the potential risk factors for its adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use Qizhi Tongluo Capsules in the monitoring hospitals.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who use Qizhi Tongluo Capsules in the monitoring hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse drug reactions (ADR) to the Qizhi Tongluo Capsules | 3 years

SECONDARY OUTCOMES:
The incidence of adverse drug event (ADE) to the Qizhi Tongluo Capsules | 3 years
The incidence of new ADRs to the Qizhi Tongluo Capsules | 3 years
The incidence of serious adverse drug event (SADE) to the Qizhi Tongluo Capsules | 3 years
Changes in biological indicators of patients with serious adverse events | 3 years
  Patients with serious adverse events and suspected unintended serious adverse reactions should be tested for liver function (ALT, AST, ALP, TBIL, DBIL)
Changes in biological indicators of patients with serious adverse events | 3 years
  Patients with serious adverse events and suspected unintended serious adverse reactions should be tested for renal function (BUN, SCr, UA)
Changes in biological indicators of patients with serious adverse events | 3 years
  Patients with serious adverse events and suspected unintended serious adverse reactions should be tested for immune indicators (IgA, IgE, T-lymphocyte, B lymphocyte, cell surface antigen, serum histamine concentration and complement).

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Ningming County Hospital of Chinese Medicine, Changzuo, Guangxi
  - Fangchenggang City Hospital of Chinese Medicine, Fangchenggang, Guangxi
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Shanglin County Hospital of Chinese Medicine, Nanning, Guangxi
  - Long'an County Hospital of Chinese Medicine, Nanning, Guangxi
  - Luohe Hospital of traditional Chinese Medicine, Luohe, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Second Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - The First Affiliated Hospital of Henan University of traditional Chinese Medicine, Zhengzhou, Henan
  - The Third Affiliated Hospital of Henan University of traditional Chinese Medicine, Zhengzhou, Henan
  - Affiliated Hospital of Yanbian University, Yanbian, Jilin
  - The Second Affiliated Hospital of Shandong University of Chinese Medicine, Jinan, Shandong
  - Affiliated Hospital of Changzhi Institute of traditional Chinese Medicine, Changzhi, Shanxi